CLINICAL TRIAL: NCT03010436
Title: The Efficacy and Safety of Benralizumab In the Treatment of Eosinophilic Grandulomatosis With Polyangiitis (EGPA) Study: BITE
Brief Title: Benralizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis (EGPA) Study
Acronym: BITE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Jewish Health (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Michael Wechsler, MD, Prinicipal Investigator, National Jewish Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3010
Record Dates: First submitted 2016-12-11; First posted 2017-01-05 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Other): All subjects will receive the study medication- benralizumab
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — one injection 30 mg under the subjects skin every 4 weeks for 8 weeks and then every 8 weeks for 24 weeks for a total of 5 treatments.

SUMMARY:
Benralizumab is a type of medicine called a monoclonal antibody that is made in the research clinic; it works by blocking a specific protein in the body called interleukin-5. The study medicine, benralizumab, is not yet approved for doctors to treat patients with EGPA. It is considered an experimental drug in this study.

DETAILED DESCRIPTION:
This study is open-label which means that all subjects will receive the study medication. The medicine-benralizumab-will be given to subjects in addition to the medicines they are already taking to treat their EGPA such as oral steroids (e.g. prednisone) and medicines that reduce the activity of their immune system. Drugs that are sometimes used (i.e., standard of care) to reduce the activity of the immune system in EGPA (in addition to oral steroids) include azathioprine, methotrexate, mycophenolate mofetil and cyclophosphamide. Information about how the stud drug that you get affects the subjects body and their health will be collected through a number of tests, procedures and questions.

The study medicine, benralizumab, will be given to subjects as one injection 30 mg under skin every four weeks for 12 weeks and then every 8 weeks for 16 weeks for a total of 5 treatments. During the treatment phase of this study, a study staff member will call the subjects to see how they are doing, what medications they are taking and if they are able to decrease their steroid use. The study is a total of 9 study visits in a 44 week time period. Everyone who takes part in the study will continue to receive his/her existing treatments for EGPA (although their dose of oral steroids may be reduced during the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Gender and Age: Male or female subjects >18 years old
* EGPA diagnosis: subjects who have been diagnosed with EGPA for at least 6 months based on the history or presence of: asthma plus eosinophilia (>1.0x109/L and/or >10% of leucocytes) plus at least two of the following additional features of EGPA

  1. A biopsy showing histopathological evidence of eosinophilic vasculitis, or perivascular eosinophilic infiltration, or eosinophil-rich granulomatous inflammation;
  2. Neuropathy, mono or poly (motor deficit or nerve conduction abnormality);
  3. Pulmonary infiltrates, non-fixed;
  4. Sino-nasal abnormality;
  5. Cardiomyopathy (established by echocardiography or MRI);
  6. Glomerulonephritis (haematuria, red cell casts, proteinuria);
  7. Alveolar haemorrhage (by bronchoalveolar lavage);
  8. Palpable purpura;
  9. ANCA positive (MPO or PR3).
* Subjects who have received cyclophosphamide can be included after a 4-week washout prior to visit 0 (first injection).
* Subjects who have received a methotrexate, azathioprine, or mycophenolate mofetil induction regimen may be included if on a stable dose for at least 4 weeks prior to visit 0.
* Corticosteroid therapy: Subject must be on a stable dose of oral prednisolone or prednisone of ≥5 mg/day for at least 4 weeks prior to visit 0.
* Immunosuppressive therapy: If receiving immunosuppressive therapy (including methotrexate, azathioprine, or mycophenolate mofetil, but excluding restricted medications below) the dosage must be stable for the 4 weeks prior to visit 0 and during the study (dose reductions for safety reasons will be permitted).
* Female subjects: Women of childbearing potential (WOCBP) must use an effective form of birth control (confirmed by the Investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective IUD intrauterine device/IUS levonogestrel Intrauterine system, Depo-Provera(tm) injections, oral contraceptive, and Evra Patch(tm) or Nuvaring(tm). WOCBP must agree to use effective method of birth control, as defined above, from enrolment, throughout the study duration and within 16 weeks after last dose of IP, and have negative serum pregnancy test result on Visit 0.
* Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of visit -1 without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
* Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
* All male subjects who are sexually active must agree to use an acceptable method of contraception (condom with or without spermicide, vasectomy) from Visit 0 until 16 weeks after their last dose.

Exclusion Criteria:

* Hypereosinophilic Syndrome
* Wegener's Granulomatosis
* History of cancer: Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent, and assent when applicable was obtained. Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent, and assent when applicable, was obtained.
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.
* Pregnant or nursing
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.5 times the upper limit of normal (ULN) confirmed during screening period.
* If female and of child-bearing potential, must have negative pregnancy test and must adhere to acceptable method of contraception (with <1% failure rate) during the study and for four months after the study.
* Receipt of any investigational non biologic within 30 days or 5 half-lives prior to visit 0, whichever is longer.
* A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
* Any other medical illness that precludes study involvement
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to be enrolled.
* Patients who are currently receiving or have previously received benralizumab or any other type of anti-interleukin therapy (i.e. mepolizumab, reslizumab, lebrikizumab etc.) within the last 4 months or 5 half-lives whichever is longer.
* History of anaphylaxis to any biologic therapy or vaccine.
* Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
* Taking cyclophosphamide

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
All adverse events will be reported by count of events (safety and tolerability ) | Up to 12 months
  All adverse events will be reported to AstraZeneca and the IRB in accordance with the policy of National Jewish Health and the FDA. Serious adverse events, whether or not considered related to the investigational drug, will be recorded on the SAE event form will be sent to AstraZeneca within 24 hours of submission to the FDA.

SECONDARY OUTCOMES:
Change in corticosteroid dosage | Up to 12 months
  Change in steroid dose will be assessed by comparing the corticosteroid dose to subjects at the end of the steroid stable phase and compare to steroid dose at the end of treatment period.
Change in the rate of EGPA exacerbations during the study period. | Up to 12 months
  Change in the rate of exacerbations will be assessed by comparing the rate of exacerbations during the study period with the rate during the washout and safety-monitoring period as well as with the self-reported rate of exacerbations from the year prior to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wechsler, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee Y, Hojjati M. Benralizumab as a Potential Adjunctive Therapy in Eosinophilic Granulomatosis With Polyangiitis. J Clin Rheumatol. 2021 Dec 1;27(8S):S401-S402. doi: 10.1097/RHU.0000000000001419. No abstract available. PMID 32453217